CLINICAL TRIAL: NCT05186610
Title: Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography and Directed Metabolic Core Needle Biopsy in the Management of Lymphoma
Brief Title: FDG PET/CT and Directed Metabolic Core Needle Biopsy in the Management of Lymphoma
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Associate Professor, Department of Nuclear Medicine,, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/1702/MD/11449-50
Record Dates: First submitted 2021-12-29; First posted 2022-01-11 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma
Keywords: Positron Emission Tomography Computed Tomography; Image-Guided Biopsy; Fluorodeoxyglucose F18; Biopsy-Core Needle
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FDG PET/CT guided metabolic core needle biopsy group: 2- Fluorodeoxyglucose (FDG) PET-positive lesions at initial presentation or at the end of treatment were considered for PET/CT guided biopsy after discussion with the hemato oncologist.
  Interventions: Procedure: FDG PET/CT guided metabolic core needle biopsy

INTERVENTIONS:
Procedure: FDG PET/CT guided metabolic core needle biopsy — The target lesion to be biopsied was chosen based on accessibility and the highest metabolic activity (Highest standardized uptake value) on FDG PET/CT imaging. The final needle course was based on the anatomic location of the lesion, FDG avidity, and its relation with vital organs. The procedures were performed under full aseptic precautions and under adequate local anesthesia. The biopsy needle was placed to the target lesion using an automated robotic arm (ARA) workstation (ROBIO-EX, Perfint healthcare Pvt Ltd, Chennai, India).

SUMMARY:
FDG-PET/CT is an established modality in various stages of management of lymphoma but definitive information regarding the diagnosis, prognostication, and further management is provided by histopathological examination. Combining the two modalities may provide an incremental benefit by identifying better sites for targetting biopsy and for better verification of sites and causes of FDG uptake seen during PET/CT.

DETAILED DESCRIPTION:
Written informed consent was obtained from all the participants for PET/CT-guided biopsy. The procedure details, related risks, and benefits were explained to all the participants. A multidisciplinary team including hemato-oncologists, nuclear medicine physicians, and pathologists were involved in the project. A hemato-oncologist decided the biopsy indication after discussing it with the nuclear medicine physician. FDG avid lesions in a clinically suspected case of lymphoma or a suspicious, residual FDG avid lesion detected at the time of follow-up PET/CT imaging in a patient with a prior diagnosis of lymphoma were sampled. The per and post-procedural complications and management were maintained in the institutional PET data registry and the final histopathological diagnosis obtained was also collected.

ELIGIBILITY:
Inclusion Criteria:

* FDG avid lesion in a clinically suspected case of lymphoma.
* Suspicious, residual FDG avid lesion detected at the time of follow-up PET/CT imaging in a patient with a prior diagnosis of lymphoma either at the end-of-treatment or during surveillance.

Exclusion Criteria:

* Deranged coagulation profile.
* Inaccessibility of the lesion for a percutaneous biopsy.
* Resolution of the lesion at the time of biopsy planning.
* Participant is not willing for the procedure.
* Pregnant females and participants less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants presenting either with clinical suspicion of lymphomatous etiology at initial documentation or follow-up PET/CT scan during interim evaluation or at the end of therapy in pathologically proven lymphomatous etiology were included. All the patients underwent whole-body FDG PET/CT imaging and the patients with a lesion suspicious for lymphomatous involvement on FDG PET/CT imaging were recruited for PET/CT guided biopsy.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The yield of FDG PET/CT guided metabolic biopsy in lymphoma | 1 year
  Percentage of biopsy procedures that yielded a sample sufficient for diagnosing the presence or absence of a specific pathology among the patients undergoing the biopsy. Negative biopsy procedures were followed up for a period of one year to confirm the negative findings.

CONTACTS AND LOCATIONS:
Overall Officials: Rajender Kumar, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Department of Nuclear Medicine, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available on reasonable request for a period of five years from the end of the study.
Supporting Information: Study Protocol
Time Frame: Five years from the end of the study period
Access Criteria: Will be made available from the principal investigator upon reasonable request.